CLINICAL TRIAL: NCT01760083
Title: A Randomized Multicentre Trial to Evaluate the Utilization of Revascularization or Optimal Medical Therapy for the Treatment of Chronic Total Coronary Occlusions
Acronym: EuroCTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Euro CTO Club (Other)
Collaborators: NHS Research and Development (Other Government); Biosensors International (Other); Asahi Intecc Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-005905-64
Record Dates: First submitted 2013-01-01; First posted 2013-01-03 (Estimated); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Chronic Stable Angina; Dyspnea; Coronary Occlusion
MeSH Terms: conditions — Angina, Stable; Dyspnea; Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biolimus-eluting stent implantation (Active Comparator): PCI of CTO using a Biomatrix drug-eluting stent system + optimal medical therapy.
  Interventions: Device: Biolimus-eluting stent implantation
- Medical therapy (No Intervention): Optimal medical therapy. Subsequent PCI only if symptoms of angina persist despite optimal medical therapy. At least 2 anti-anginal agents or the maximum tolerated anti-anginal therapy should be used before crossover. Medical therapy should include adequate ventricular rate-limiting medication (i.e. Beta-blocker or rate-limiting calcium antagonist) where appropriate.

INTERVENTIONS:
Device: Biolimus-eluting stent implantation — Recanalization of chronic coronary artery occlusion and subsequent implantation of one or ore Biosensor stents
  Other Names: Biosensors Biolimus-eluting stents of all sizes and lengths
  Arms: Biolimus-eluting stent implantation

SUMMARY:
CTOs are common among patients with angina, and are detected in around 20% of patients undergoing coronary angiography. Treatment of CTO has been found to constitute only 7% of PCI practice on average. One of the reasons for the under-presentation of CTOs in PCI target lesions is the lack of evidence-based medical data on treatment indications, and the continued low level of accepted evidence for the treatment of CTOs by PCI in PCI guidelines.

Patients with a CTO represent patients with stable coronary artery disease. The COURAGE trial comparing PCI with optimal medical therapy in stable coronary disease did not show a difference in mortality or myocardial infarction between the two treatment options. However, CTOs were not included in the COURAGE trial. But that trial did confirm the superiority of PCI over OMT in controlling symptoms of angina, with a high cross-over rate to PCI. Whether PCI for CTO is superior to OMT in reducing MACE in those patients with a large ischaemic burden has never been tested in a randomized controlled trial.

While there is compelling evidence from registry studies of a clinical and prognostic benefit following successful PCI of CTO compared with PCI failure, there has been no randomized controlled trial of contemporary PCI using drug-eluting stents versus optimal medical therapy. The COURAGE trial nuclear sub-study confirms both that prognosis is closely related to the extent of residual ischaemia and that PCI is more effective in reducing residual ischaemia than optimal medical therapy alone. This confirms earlier retrospective data suggesting that the benefit of PCI is greatest in patients with moderate (10-20%) or severe (>20%) ischaemia.

Study hypothesis: PCI with Biolimus eluting stent implantation plus OMT will be superior to OMT alone in improving health status at 12-month follow-up, and will be noninferior with respect to the composite of all cause death/ non fatal MI at 36-month follow up, in patients with a CTO in an epicardial coronary artery >2.5 mm diameter and chronic stable angina with evidence of ischemia and viability in the territory subtended by the CTO

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age with written informed consent
* CTO in native coronary artery
* a) Stable angina, or b) myocardial ischaemia in a territory supplied by CTO, and c) viability in akinetic myocardium (<50% transmural late enhancement on MRI or normal resting perfusion scan)
* CTO located in segments 1-3 (RCA), 6-7 (LAD), 11-12 (LCx)
* target artery ≥2.5mm

Exclusion Criteria:

* AMI or NSTE-ACS within 1 month
* Significant untreated coronary stenosis in a territory other than CTO
* Patients with MVD and significant non-CTO stenoses where it is deemed unsafe to treat the non-CTO lesion first (e.g. Significant proximal LAD lesion with chronically occluded RCA)
* Patient unsuitable for 12 month dual anti-platelet therapy
* Any exclusion criteria for PCI or DES
* Pregnant or nursing patients and those who plan pregnancy in the period up to 1 year following index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Quality of Life Seattle Angina Questionnaire (SAQ) | Baseline and 12 months
  Seattle Angina Questionnaire and EQ-5D for health outcomes measurement
Major cardiovascular events | 36 months
  Cumulative composite endpoint of cardiovascular death, non-fatal MI at 3 years

SECONDARY OUTCOMES:
Safety and efficacy endpoints | 12 and 36 months
  All cause mortality Cardiac mortality Myocardial Infarction Any hospitalization due to cardiovascular events (angina, congestive heart failure, arrythmias) Repeat revascularization
Procedural complications | baseline upto 36 months
  Incl. periprocedural enzyme leak (defined by CK increase >3 times ULN); pericprocedural MI (new Q-wave or STEMI); pericardial tamponade, need for urgent CABG, CIN, death within 30 days, proven periprocedural cerebrovascular events
Protocol adherence | 36 months
  Need to cross from OMT to PCI in Group 2 (after escalation up to maximum tolerated anti-anginal therapy and persistent unequivocal symptoms)
Per protocol analysis | 36 months
  primary endpoint comparison in patients who did have a successful revascularization compared to those patients treated medically who had no subsequent PCI

OTHER OUTCOMES:
Health-economic analysis | 12 and 36 months
  Economic assessment & cost efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Gerald S Werner, MD PhD, Principal Investigator — Klinikum Darmstadt, Darmstadt Germany
Locations (19):
- France (5):
  - Clinique Saint-Augustin, Bordeaux
  - CH de Lagny, Lagny
  - Institut Hospitalier Jacques Cartier - ICPS, Massy
  - Clinique Pasteur, Toulouse
  - Rangueil university hospital, Toulouse
- Germany (4):
  - Zentralklinik Bad Berka, Bad Berka
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Main Taunus Kliniken, Bad Soden
  - Klinikum Darmstadt, Darmstadt
- Cardiac Catheterization Laboratory and Cardiovascular Interventional Unit Cannizzaro Hospita, Catania, Italy
- Latvian Center of Cardiology Pauls Stradins Clinical University Hospital, Riga, Latvia
- Spain (4):
  - Unidad de Cardiología Intervencionista Hospital de Sant Pau, Barcelona
  - Hospital Clinic Villaroel, Barcelona
  - Hospital Galdakao-Usansolo, Galdakao
  - Cardiovascular Institute - Hospital Clinico San Carlos, Madrid
- United Kingdom (4):
  - Royal Sussex County Hospital - Brighton and Sussex University Hospitals, Brighton
  - Royal Infirmary of Edinburgh, Edinburgh
  - Department of Cardiovascular Sciences University of Leicester, Leicester
  - National Heart and Lung Institute Imperial College, London

REFERENCES:
- [Result] Werner GS, Martin-Yuste V, Hildick-Smith D, Boudou N, Sianos G, Gelev V, Rumoroso JR, Erglis A, Christiansen EH, Escaned J, di Mario C, Hovasse T, Teruel L, Bufe A, Lauer B, Bogaerts K, Goicolea J, Spratt JC, Gershlick AH, Galassi AR, Louvard Y; EUROCTO trial investigators. A randomized multicentre trial to compare revascularization with optimal medical therapy for the treatment of chronic total coronary occlusions. Eur Heart J. 2018 Jul 7;39(26):2484-2493. doi: 10.1093/eurheartj/ehy220. PMID 29722796
- [Derived] Werner GS, Hildick-Smith D, Martin Yuste V, Boudou N, Sianos G, Gelev V, Rumoroso JR, Erglis A, Christiansen EH, Escaned J, Di Mario C, Teruel L, Bufe A, Lauer B, Galassi AR, Louvard Y. Three-year outcomes of A Randomized Multicentre Trial Comparing Revascularization and Optimal Medical Therapy for Chronic Total Coronary Occlusions (EuroCTO). EuroIntervention. 2023 Sep 18;19(7):571-579. doi: 10.4244/EIJ-D-23-00312. PMID 37482940
- [Derived] Azzalini L, Vo M, Dens J, Agostoni P. Myths to Debunk to Improve Management, Referral, and Outcomes in Patients With Chronic Total Occlusion of an Epicardial Coronary Artery. Am J Cardiol. 2015 Dec 1;116(11):1774-80. doi: 10.1016/j.amjcard.2015.08.050. Epub 2015 Sep 11. PMID 26434510
- See also: Sponsor European CTO Club e.V. (ECC) — http://eurocto.eu